CLINICAL TRIAL: NCT06876454
Title: Optimal Nutritional Palliation of Obstructed GEJ Cancer
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Responsible Party: Principal Investigator, Rahul Nayak, Director of Research, London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Nutrition Palliation of GEJ Ca
Record Dates: First submitted 2025-03-10; First posted 2025-03-14 (Actual); Last update posted 2025-05-25 (Actual); Status verified 2025-03

CONDITIONS: Esophageal Cancer
Keywords: metastatic; obstructing
MeSH Terms: conditions — Esophageal Neoplasms; Neoplasm Metastasis

STUDY DESIGN:
Intervention Model Description: This study is a single centre, prospective, feasibility randomized controlled clinical trial.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Gastrostomy Tube (Active Comparator): Gastrostomy Tube insertion for palliation
  Interventions: Procedure: Gastrostomy Tube
- Esophageal Stent (Active Comparator): Self Expanding Esophageal stent insertion for palliation
  Interventions: Device: Self Expanding Metal esophageal Stent

INTERVENTIONS:
Procedure: Gastrostomy Tube — Feeding gastrostomy tube insertion
  Arms: Gastrostomy Tube
Device: Self Expanding Metal esophageal Stent — Fully covered SEMS in the esophagus
  Arms: Esophageal Stent

SUMMARY:
The main goal of this trial is to assess whether it's feasible to conduct a larger, full-scale study comparing the use of gastrostomy (g-tubes) and stents in patients with unresectable cancer of the stomach and/or esophagus, and to evaluate their impact on patients' quality of life. Additional objectives include examining the rates of complications, the need for additional treatments, and the total number of hospital days over a three-month period.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18 years of age and older who present with an obstructing metastatic or unresectable gastroesophageal cancer.

Exclusion Criteria:

* Patients under the age of 18 years.
* Prior Esophageal Stent or gastrostomy tube

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Estimated)
Dates: Start 2025-07-01 (Estimated); Primary Completion 2026-07-01 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
FACT-E | 3 months
  • Change in FACT-E scores

SECONDARY OUTCOMES:
Complications | 3 months
  • The rates of grade 1 to 5 complications as per the TSQIC
Crossover | 3 months
  Rate of crossover from initial intervention to comparator arm

CONTACTS AND LOCATIONS:
Overall Officials: Rahul Nayak, MD MSc, Principal Investigator — London Health Sciences Centre
Locations (1):
- London Health Sciences Centre - Victoria Hospital, London, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Yes
age, date of death, intervention received, complications from intervention, FACT-E score will be available as supplemental data in the final publication. A master list will be kept on site and can be shared if there are other collaborative projects and/or a data audit is required to validate final results.
Supporting Information: Study Protocol, SAP, CSR

REFERENCES:
- [Background] Brenner DR, Weir HK, Demers AA, Ellison LF, Louzado C, Shaw A, Turner D, Woods RR, Smith LM; Canadian Cancer Statistics Advisory Committee. Projected estimates of cancer in Canada in 2020. CMAJ. 2020 Mar 2;192(9):E199-E205. doi: 10.1503/cmaj.191292. Epub 2020 Mar 2. PMID 32122974
- [Background] Kakuta T, Kosugi SI, Ichikawa H, Hanyu T, Ishikawa T, Kanda T, Wakai T. Palliative interventions for patients with incurable locally advanced or metastatic thoracic esophageal carcinoma. Esophagus. 2019 Jul;16(3):278-284. doi: 10.1007/s10388-019-00665-0. Epub 2019 Apr 4. PMID 30949884
- [Background] Philips P, North DA, Scoggins C, Schlegel M, Martin RC. Gastric-Esophageal Stenting for Malignant Dysphagia: Results of Prospective Clinical Trial Evaluation of Long-Term Gastroesophageal Reflux and Quality of Life-Related Symptoms. J Am Coll Surg. 2015 Jul;221(1):165-73. doi: 10.1016/j.jamcollsurg.2015.01.062. Epub 2015 Feb 28. PMID 26095567
- [Background] Yu FJ, Shih HY, Wu CY, Chuang YS, Lee JY, Li HP, Fang PT, Tsai DL, Chou SH, Wu IC. Enteral nutrition and quality of life in patients undergoing chemoradiotherapy for esophageal carcinoma: a comparison of nasogastric tube, esophageal stent, and ostomy tube feeding. Gastrointest Endosc. 2018 Jul;88(1):21-31.e4. doi: 10.1016/j.gie.2017.11.030. Epub 2017 Dec 7. PMID 29225081
- [Background] Madhusudhan C, Saluja SS, Pal S, Ahuja V, Saran P, Dash NR, Sahni P, Chattopadhyay TK. Palliative stenting for relief of dysphagia in patients with inoperable esophageal cancer: impact on quality of life. Dis Esophagus. 2009;22(4):331-6. doi: 10.1111/j.1442-2050.2008.00906.x. PMID 19473211
- [Background] Amin S, Lin C. Immunotherapy Plus Chemoradiation Improves Overall Survival in Stage IV Esophageal Cancer: A Cohort Study. Gastro Hep Adv. 2023 Dec 12;3(3):302-310. doi: 10.1016/j.gastha.2023.12.004. eCollection 2024. PMID 39131143